CLINICAL TRIAL: NCT06488092
Title: Implementation of Calculated Cesarean Section Risk Study: Patient-focused Outcomes
Brief Title: IC-CS Risk: Patient Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rebecca Feldman Hamm, Assistant Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 854955
Record Dates: First submitted 2024-06-25; First posted 2024-07-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Delivery

STUDY DESIGN:
Intervention Model Description: This is a quality improvement randomized roll-out pre-implementation and post-implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-utilization of cesarean risk calculator (No Intervention): The time prior to the implementation of the cesarean risk calculator at the labor and delivery unit.
- Implementation of cesarean risk calculator (Active Comparator): The cesarean risk calculator will be incorporated into routine care at the site
  Interventions: Other: Cesarean Risk Calculator

INTERVENTIONS:
Other: Cesarean Risk Calculator — The cesarean risk calculator will be incorporated into routine care at the site
  Arms: Implementation of cesarean risk calculator

SUMMARY:
This study is looking at the impact of the implementation of a cesarean risk calculator on cesarean delivery and maternal morbidity rates.

DETAILED DESCRIPTION:
In this study a cesarean risk calculator will be instituted as a part of standard of care in a randomized rollout at 14 labor and delivery clinical sites across 4 institutions. The leadership at all of the sites have planned to implement this intervention for routine use at both sites. This study will evaluate cesarean delivery rates and maternal morbidity before and after implementation at each site.

ELIGIBILITY:
Inclusion Criteria:

All postpartum patients who were eligible for cesarean risk calculator utilization:

* delivery of a full-term (greater than or equal to 37 weeks) singleton gestation after presenting
* with intact membranes
* undergoing an induction of labor from cervical dilation less than or equal to 2cm

Exclusion Criteria:

Postpartum patient who had a prior pregnancy resulting in Cesarean delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Cesarean delivery rate (for any indication) | at time of delivery
Maternal morbidity | from delivery to 30 days postpartum
  one or more of the following: endometritis, postpartum hemorrhage greater than or equal to one liter, wound infection requiring antibiotics, venous thromboembolism, hysterectomy, intensive care unit admission, readmission within 30 days, and death

SECONDARY OUTCOMES:
Neonatal morbidity | delivery admission
  one or more of the following: severe respiratory distress, neonatal resuscitation outside of delivery room, and sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hamm, MD, Principal Investigator — University of Pennsylvania
Locations (14):
- United States (14):
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - E.W. Sparrow Hospital, Lansing, Michigan
  - Princeton Medical Center, Plainsboro, New Jersey
  - Akron General, Akron, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Lancaster General Health, Lancaster, Pennsylvania
  - Chester County Hosptial, West Chester, Pennsylvania
  - Logan Regional Hospital-Intermountain Healthcare, Logan, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Riverton Hospital-Intermountain Healthcare, Riverton, Utah
  - University of Utah Hospital, Salt Lake City, Utah